CLINICAL TRIAL: NCT02765269
Title: Development and Testing of an Intelligent Pain Management System (IPMS) for Chinese Patients With Cancer
Brief Title: Intelligent Pain Management System for Assessing Pain in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Translational Institute for Cancer Pain, Shanghai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: XHTICP 001
Record Dates: First submitted 2016-04-25; First posted 2016-05-06 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-07

CONDITIONS: Pain; Neoplasms
Keywords: cancer pain; mobile applications
MeSH Terms: conditions — Pain; Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPMS group (Experimental): Cancer patients with pain are asked to use the Intelligent Pain Management System as much as possible to record the degree and location of pain at least once every day. Through assessments of these pain record, physicians could give the patients appropriate advice.
  Interventions: Device: Intelligent Pain Management System
- Control group (No Intervention): The control group are communicated through conventional method such as telephone calls or door-to-door visit to collect the pain assessment to guide doctors' therapy.

INTERVENTIONS:
Device: Intelligent Pain Management System — A mobile phone application which can record the pain the cancer patients have and can deliver these records to doctors in order that doctors give patients prescriptions promptly.
  Other Names: IPMS
  Arms: IPMS group

SUMMARY:
The purpose of this study is to determine whether the Intelligent Pain Management System (IPMS) could make recording and interfering pain timely among cancer patients with pain. The system's usability, feasibility, compliance, and satisfaction will also be assessed.

DETAILED DESCRIPTION:
Research indicate that over one-third of cancer patients experienced cancer pain, which is known as a major reason leading to lower quality of life of the patients.In this present study, the investigators aim to design, develop, and test the feasibility of a low cost, conveniently implemented mobile application to facilitate real-time pain recording and timely intervention among Chinese cancer patients with pain. This system evaluate real-time pain and Karnofsky Performance Status（KPS）scores for quality of life, and to generate an action plan to visit the physician or to adjust pain medication dosage when the pain threshold is reached. The investigators study is to test this system's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* the patient was able to read Chinese and use smart phones;
* the patient was diagnosed with cancer and has self-reported cancer pain within a month prior to the study;
* the patient was being seen on a regular basis by the oncology team;
* the patient was under standard analgesia treatments;
* the patient was estimated to have over 3 months survival time.

Exclusion Criteria:

* the patients who self-reported to have severe cognitive impairments or major comorbid illnesses that would interfere with pain assessment.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Ding, Study Chair — Xinhua Hospital Affliated to Shanghai Jiao Tong University School of Medicine, Chongming Branch
Locations (1):
- Xinhua Translational Institute for Cancer Pain, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun Y, Jiang F, Gu JJ, Wang YK, Hua H, Li J, Cheng Z, Liao Z, Huang Q, Hu W, Ding G. Development and Testing of an Intelligent Pain Management System (IPMS) on Mobile Phones Through a Randomized Trial Among Chinese Cancer Patients: A New Approach in Cancer Pain Management. JMIR Mhealth Uhealth. 2017 Jul 25;5(7):e108. doi: 10.2196/mhealth.7178. PMID 28743681

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IPMS Group | Control Group
Started | 25 | 21
Completed | 25 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPMS Group | Control Group | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 15 | 15 | 30
Gender [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 19 | 13 | 32
Region of Enrollment [Number; unit: participants]
  China | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Mobile Application Assessed by Observing the Number of Daily Pain Assessments Recorded Among Patients
Description: The primary objective is to demonstrate that this mobile application is feasible by observing the numbers of daily pain assessment among patients.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: pain assessments per day
Arm/Group | IPMS Group | Control Group
Number analyzed (Participants) | 25 | 0
pain assessments per day | 2.37 (0.53) |

2. Secondary Outcome: Pain Management
Description: Numerical rating scale allows a person to describe the intensity of his/her pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be". Higher values means worse outcomes. The investigators will compare average pain score assessed by numerical rating scale at the end of the trial period.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IPMS Group | Control Group
Number analyzed (Participants) | 25 | 21
scores on a scale | 2.20 (0.50) | 2.95 (0.59)

3. Secondary Outcome: Users' Satisfaction (Questionnaire)
Description: Patients will be asked to complete a questionnaire after patients use it for 2 weeks.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | IPMS Group | Control Group
Number analyzed (Participants) | 25 | 0
participants
  very much like IPMS | 9 |
  like IMPS | 16 |
  dislike IPMS | 0 |

4. Secondary Outcome: Karnofsky Performance Score Evaluation
Description: The Karnofsky performance score runs from 100 to 0, where 100 is "perfect" health and 0 is death. Higher values represent better outcomes.The investigators will compare average score between trial group and control group.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IPMS Group | Control Group
Number analyzed (Participants) | 25 | 21
scores on a scale | 68.80 (7.23) | 56.19 (7.40)

ADVERSE EVENTS:
Description: No adverse events were assessed throughout the study.
Arm/Group | IPMS Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes